CLINICAL TRIAL: NCT03139383
Title: Intraoperative Intravenous Dextrose Administration and the Incidence of Nausea and Vomiting After the Gynecologic Laparoscopic Surgery A Randomized Double-Blinded Controlled Study
Brief Title: Dextrose Containing Fluid and the Postoperative Nausea and Vomiting in the Gynecologic Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Pathomporn Pin on, M.D., Assistant professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANE-2557-02323; 2519-04-17 (Other: Asian Biomedicine)
Record Dates: First submitted 2017-04-30; First posted 2017-05-04 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: postoperative nausea; postoperative vomiting; gynecologic laparoscopic surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Glucose; Saline Solution

STUDY DESIGN:
Intervention Model Description: a prospective randomized double-blind controlled study of the incidence and severity of postoperative nausea and vomiting in female participants receiving different types of intravenous fluid solution
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients did not know the type of intravenous fluid they received during the surgery. The outcome assessors were blineded too.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal saline solution (Placebo Comparator): The patients received normal saline solution as a maintenance fluid during surgery in dose of 2 ml/kg/hour.
  Interventions: Other: saline solution
- dextrose solution (Active Comparator): The patients received dextrose solution as a maintenance fluid during surgery in dose of 2 ml/kg/hour.
  Interventions: Other: dextrose solution

INTERVENTIONS:
Other: dextrose solution — The patients received 5%D/N/2 during surgery
  Other Names: 5% dextrose in half strength saline solution
  Arms: dextrose solution
Other: saline solution — The patients received NSS during surgery
  Other Names: normal saline solution
  Arms: normal saline solution

SUMMARY:
The investigators tested the hypothesis that administration of intravenous dextrose as a maintenance fluid in gynecologic laparoscopic surgery would reduce the incidence and severity of postoperative nausea and vomiting (PONV) compared with normal saline solution in the same dose.

A prospective randomized double blinded controlled study was conducted. Eighty six participants were randomized to dextrose solution (n= 42) or normal saline solution (n= 44). The Bellville postoperative nausea and vomiting scores were recorded until 24 hours after surgery.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a major complication in laparoscopic gynecologic surgery. There are limited data and conflicting results from previous studies related to the types of intravenous fluid and a reduction in PONV. The incidence of nausea is slightly greater than the incidence of vomiting (50% vs. 30%). General anesthesia increased the likelihood of PONV 11 times compared with other types of anesthesia. Laparoscopic surgery can further increase the incidence of PONV to 80%.Identified risk factors of PONV included female, history of motion sickness, nonsmoking, younger age, general anesthesia, use of volatile anesthetics and nitrous oxide, opioids, duration of anesthesia, and types of surgery (cholecystectomy, laparoscopic, gynecological). Adequate intravenous fluid hydration is another effective strategy for reducing the baseline risk for PONV (Evidence A2). Previous studies showed that there was no difference in efficacy between crystalloids and colloids when similar volumes were used in surgeries associated with minimal fluid shifts. While liberal intravenous fluid administration, such as 30 ml/ kg of sodium lactate solution, reduced the incidence of PONV after gynecologic laparoscopy compared to another group receiving 10 ml/kg of sodium lactate solution, this strategy did not reduce the PONV in other surgical procedures such as thyroidectomy. Among crystalloid solutions, results from previous studies were conflicting regarding the benefit of intravenous dextrose administration to reducing the PONV. Hypovolemia with and without hypoglycemia after overnight fasting were believed to exacerbate PONV.

The investigators hypothesized that intraoperative infusion of dextrose solution could reduce the incidence and severity of PONV. The investigators proposed to determine the relationship between types of fluid administration and antiemetic requirement and serum glucose in paricipants scheduled for the gynecologic laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* elective surgery
* Gynecologic laparoscopic surgery
* give informed consent

Exclusion Criteria:

* pregnancy
* DM
* congestive heart failure

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — the surgical procedure was done only in female patients
Enrollment: 100 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2015-09-28 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
the incidence and severity of postoperative nausea and vomiting | 24 hour after surgery
  Bellville score assessment

SECONDARY OUTCOMES:
Antiemetic drug requirement | 24 hour after surgery
  nausea and vomiting drugs requested by the patients
serum glucose | 2 hour after surgery
  DTX was assessed

CONTACTS AND LOCATIONS:
Overall Officials: Pathomporn Pin-on, Principal Investigator — Chiang Mai University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinclair DR, Chung F, Mezei G. Can postoperative nausea and vomiting be predicted? Anesthesiology. 1999 Jul;91(1):109-18. doi: 10.1097/00000542-199907000-00018. PMID 10422935
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Koivuranta M, Laara E, Snare L, Alahuhta S. A survey of postoperative nausea and vomiting. Anaesthesia. 1997 May;52(5):443-9. doi: 10.1111/j.1365-2044.1997.117-az0113.x. PMID 9165963
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162